CLINICAL TRIAL: NCT03083834
Title: Salivary Free Cortisol Response to Cosyntropin Stimulation Test in Mitotane Treated Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, leonard.saiegh, MD, Bnai Zion Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0006-17-BNZ
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Adrenal Insufficiency; Adrenal Cancer
Keywords: cosyntropin; salivary free cortisol; mitotane
MeSH Terms: conditions — Adrenal Insufficiency; Adrenal Gland Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- healthy subjects (Experimental): low-dose cosyntropin stimulation test
  Interventions: Diagnostic Test: Cosyntropin stimulation test
- hypoadrenal mitotane treated patients (Experimental): low-dose cosyntropin stimulation test
  Interventions: Diagnostic Test: Cosyntropin stimulation test
- hypoadrenal no-mitotane treated patients (Experimental): low-dose cosyntropin stimulation test
  Interventions: Diagnostic Test: Cosyntropin stimulation test

INTERVENTIONS:
Diagnostic Test: Cosyntropin stimulation test — At 0800h to 0900h, a 25 mm plastic intravenous line will be inserted in an antecubital vein. Then, 1 μg/ml ACTH aliquot stock solution will be pushed through, followed by 5 ml physiologic saline (0.9%). Serum cortisol and salivary free cortisol will measured just before ACTH administration and 30 minutes later.

SUMMARY:
In mitotane treated patients, serum cortisol cannot be used to diagnose hypoadrenalism, since mitotane increases cortisol binding globulin levels (CBG), artificially raising total cortisol. Salivary free cortisol (SC) is not affected by CBG alterations, and reflects the free serum cortisol.

In the current study, investigators will assess serum and SC responses during low-dose cosyntropin stimulation test in healthy volunteers, mitotane-induced hypoadrenal patients on steroid replacement therapy and in patients who suffer from hypoadrenlism caused from other etiology. Investigators will compare results between groups and try to demonstrate the superiority of SC in assessing adrenal function in mitotane treated patients.

DETAILED DESCRIPTION:
80-90% of circulating cortisol is bound to cortisol binding globulin (CBG) or transcortin, whereas only 3-10% is in the free state. Salivary free cortisol (SC) is an index of plasma free cortisol. In previous studies it was shown that in low-dose cosyntropin stimulation test, SC increases significantly in normal but not in hypoadrenal patients. It was suggested that dynamic assessment of the SC response to ACTH may be particularly helpful whenever the measurement of serum cortisol is complicated by increased or decreased CBG levels.

Adrenocortical carcinoma (ACC) is a rare malignancy with a heterogeneous presentation and a variable but generally poor prognosis. Mitotane is the main drug for ACC treatment and it plays a role both in adjuvant treatment after complete resection and in recurrent, inoperable and/or metastatic ACC. Mitotane blocks adrenocortical steroid synthesis and also exerts a specific cytotoxic effect on adrenocortical cells. Mitotane induces adrenal insufficiency, requiring hydrocortisone replacement therapy. In mitotane treated patients, serum cortisol cannot be used to diagnose hypoadrenalism, since mitotane increases CBG levels, artificially raising total cortisol. SC is not affected by CBG alterations, and reflects the free serum cortisol and may be more accurate in diagnosing hypoadrenalism in mitotane treated patients.

In the current study, investigators will assess serum and SC responses during low-dose cosyntropin stimulation test in healthy volunteers, mitotane-induced hypoadrenal patients on steroid replacement therapy and in patients who suffer from hypoadrenlism caused from any other etiology. Investigators will compare results between groups and try to demonstrate the superiority of SC in assessing adrenal function in mitotane treated patients.

ELIGIBILITY:
Inclusion Criteria:

* mitotane treated
* known hypoadrenlism

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-03-14 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Salivary free cortisol | 1 day
  Salivary free cortisol concentrations during intravenous low dose cosyntropin stimulation test..

SECONDARY OUTCOMES:
serum cortisol | 1 day
  Serum cortisol concentrations during intravenous low dose cosyntropin stimulation test.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Saiegh, MD, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bnai Zion MC, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No